CLINICAL TRIAL: NCT00783887
Title: Molecular Diagnosis of Primary Ciliary Dyskinesia
Brief Title: Diagnosis of Primary Ciliary Dyskinesia
Acronym: DCP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 06053
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
Keywords: Cilia; Axoneme; Dynein; Gene; Ultrastructure; Linkage analysis
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, Serum, White blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with suspected or confirmed primary ciliary dyskinesia after ciliary investigations who accepted to participate to the genetic studies
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample of 5 ml

SUMMARY:
Primary ciliary dyskinesia is an inherited respiratory disease caused by various functional and ultrastructural abnormalities of respiratory cilia. The genetic heterogeneity underlying PCD is extremely important and only few genes are clearly implicated in PCD. Their mutations account for about 20% of patients. For all the other PCD patients, the genes responsible for their ciliary defect remain to be identify.

DETAILED DESCRIPTION:
1/ Evaluating the frequency of mutations of the two main genes implicated in PCD, in a large cohort of patients with PCD confirmed by ciliary investigations.2/ Identifying and testing new candidate genes responsible not only for typical PCD and related disorders of the axoneme, but also for so far-unexplored "syndromic forms of PCD", taking advantage of data obtained through comparative genomic approaches between different species, ciliated or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or confirmed primary ciliary dyskinesia after ciliary investigations who accepted to participate to the genetic studies.

Exclusion Criteria:

* Patients with exclusion of primary ciliary dyskinesia after ciliary investigations.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected or confirmed primary ciliary dyskinesia (followed by the participating centers)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
After DNA extraction,standard procedures for the identification of human gene mutations will be used for each gene tested in the study | At the inclusion visit

SECONDARY OUTCOMES:
Complementary ciliary investigations in patients with suspected primary ciliary dyskinesia. | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Serge AMSELEM, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital A. Trousseau, Service de Génétique et d'Embryologie Médicales, Paris, France

REFERENCES:
- [Background] Bush A, Cole P, Hariri M, Mackay I, Phillips G, O'Callaghan C, Wilson R, Warner JO. Primary ciliary dyskinesia: diagnosis and standards of care. Eur Respir J. 1998 Oct;12(4):982-8. doi: 10.1183/09031936.98.12040982. PMID 9817179
- [Background] Noone PG, Leigh MW, Sannuti A, Minnix SL, Carson JL, Hazucha M, Zariwala MA, Knowles MR. Primary ciliary dyskinesia: diagnostic and phenotypic features. Am J Respir Crit Care Med. 2004 Feb 15;169(4):459-67. doi: 10.1164/rccm.200303-365OC. Epub 2003 Dec 4. PMID 14656747
- [Background] Holzmann D, Ott PM, Felix H. Diagnostic approach to primary ciliary dyskinesia: a review. Eur J Pediatr. 2000 Jan-Feb;159(1-2):95-8. doi: 10.1007/pl00013813. PMID 10653339
- [Background] Afzelius BA, Gargani G, Romano C. Abnormal length of cilia as a possible cause of defective mucociliary clearance. Eur J Respir Dis. 1985 Mar;66(3):173-80. PMID 3979484
- [Background] Escudier E, Escalier D, Pinchon MC, Boucherat M, Bernaudin JF, Fleury-Feith J. Dissimilar expression of axonemal anomalies in respiratory cilia and sperm flagella in infertile men. Am Rev Respir Dis. 1990 Sep;142(3):674-9. doi: 10.1164/ajrccm/142.3.674. PMID 2389919
- [Background] Verra F, Fleury-Feith J, Boucherat M, Pinchon MC, Bignon J, Escudier E. Do nasal ciliary changes reflect bronchial changes? An ultrastructural study. Am Rev Respir Dis. 1993 Apr;147(4):908-13. doi: 10.1164/ajrccm/147.4.908. PMID 8466127
- [Background] Wodehouse T, Kharitonov SA, Mackay IS, Barnes PJ, Wilson R, Cole PJ. Nasal nitric oxide measurements for the screening of primary ciliary dyskinesia. Eur Respir J. 2003 Jan;21(1):43-7. doi: 10.1183/09031936.03.00305503. PMID 12570107
- [Background] Arnal JF, Flores P, Rami J, Murris-Espin M, Bremont F, Pasto I Aguilla M, Serrano E, Didier A. Nasal nitric oxide concentration in paranasal sinus inflammatory diseases. Eur Respir J. 1999 Feb;13(2):307-12. doi: 10.1034/j.1399-3003.1999.13b15.x. PMID 10065673
- [Background] Karadag B, James AJ, Gultekin E, Wilson NM, Bush A. Nasal and lower airway level of nitric oxide in children with primary ciliary dyskinesia. Eur Respir J. 1999 Jun;13(6):1402-5. doi: 10.1183/09031936.99.13614069. PMID 10445619
- [Background] Rossman CM, Lee RM, Forrest JB, Newhouse MT. Nasal cilia in normal man, primary ciliary dyskinesia and other respiratory diseases: analysis of motility and ultrastructure. Eur J Respir Dis Suppl. 1983;127:64-70. PMID 6225660
- [Background] Chilvers MA, Rutman A, O'Callaghan C. Functional analysis of cilia and ciliated epithelial ultrastructure in healthy children and young adults. Thorax. 2003 Apr;58(4):333-8. doi: 10.1136/thorax.58.4.333. PMID 12668798
- [Background] Tamalet A, Clement A, Roudot-Thoraval F, Desmarquest P, Roger G, Boule M, Millepied MC, Baculard TA, Escudier E. Abnormal central complex is a marker of severity in the presence of partial ciliary defect. Pediatrics. 2001 Nov;108(5):E86. doi: 10.1542/peds.108.5.e86. PMID 11694670
- [Background] Moore A, Escudier E, Roger G, Tamalet A, Pelosse B, Marlin S, Clement A, Geremek M, Delaisi B, Bridoux AM, Coste A, Witt M, Duriez B, Amselem S. RPGR is mutated in patients with a complex X linked phenotype combining primary ciliary dyskinesia and retinitis pigmentosa. J Med Genet. 2006 Apr;43(4):326-33. doi: 10.1136/jmg.2005.034868. Epub 2005 Jul 31. PMID 16055928
- [Background] Krawczynski MR, Witt M. PCD and RP: X-linked inheritance of both disorders? Pediatr Pulmonol. 2004 Jul;38(1):88-9. doi: 10.1002/ppul.30001. PMID 15170879
- [Background] Pennarun G, Escudier E, Chapelin C, Bridoux AM, Cacheux V, Roger G, Clement A, Goossens M, Amselem S, Duriez B. Loss-of-function mutations in a human gene related to Chlamydomonas reinhardtii dynein IC78 result in primary ciliary dyskinesia. Am J Hum Genet. 1999 Dec;65(6):1508-19. doi: 10.1086/302683. PMID 10577904
- [Background] Porter ME. Axonemal dyneins: assembly, organization, and regulation. Curr Opin Cell Biol. 1996 Feb;8(1):10-7. doi: 10.1016/s0955-0674(96)80042-1. PMID 8791407
- [Background] Porter ME, Sale WS. The 9 + 2 axoneme anchors multiple inner arm dyneins and a network of kinases and phosphatases that control motility. J Cell Biol. 2000 Nov 27;151(5):F37-42. doi: 10.1083/jcb.151.5.f37. No abstract available. PMID 11086017
- [Background] Zariwala M, Noone PG, Sannuti A, Minnix S, Zhou Z, Leigh MW, Hazucha M, Carson JL, Knowles MR. Germline mutations in an intermediate chain dynein cause primary ciliary dyskinesia. Am J Respir Cell Mol Biol. 2001 Nov;25(5):577-83. doi: 10.1165/ajrcmb.25.5.4619. PMID 11713099
- [Background] Guichard C, Harricane MC, Lafitte JJ, Godard P, Zaegel M, Tack V, Lalau G, Bouvagnet P. Axonemal dynein intermediate-chain gene (DNAI1) mutations result in situs inversus and primary ciliary dyskinesia (Kartagener syndrome). Am J Hum Genet. 2001 Apr;68(4):1030-5. doi: 10.1086/319511. Epub 2001 Feb 23. PMID 11231901
- [Background] Dutcher SK. Chlamydomonas reinhardtii: biological rationale for genomics. J Eukaryot Microbiol. 2000 Jul-Aug;47(4):340-9. doi: 10.1111/j.1550-7408.2000.tb00059.x. PMID 11140447
- [Background] Kamiya R. Functional diversity of axonemal dyneins as studied in Chlamydomonas mutants. Int Rev Cytol. 2002;219:115-55. doi: 10.1016/s0074-7696(02)19012-7. PMID 12211628
- [Background] Pennarun G, Chapelin C, Escudier E, Bridoux AM, Dastot F, Cacheux V, Goossens M, Amselem S, Duriez B. The human dynein intermediate chain 2 gene (DNAI2): cloning, mapping, expression pattern, and evaluation as a candidate for primary ciliary dyskinesia. Hum Genet. 2000 Dec;107(6):642-9. doi: 10.1007/s004390000427. PMID 11153919
- [Background] Bartoloni L, Blouin JL, Maiti AK, Sainsbury A, Rossier C, Gehrig C, She JX, Marron MP, Lander ES, Meeks M, Chung E, Armengot M, Jorissen M, Scott HS, Delozier-Blanchet CD, Gardiner RM, Antonarakis SE. Axonemal beta heavy chain dynein DNAH9: cDNA sequence, genomic structure, and investigation of its role in primary ciliary dyskinesia. Genomics. 2001 Feb 15;72(1):21-33. doi: 10.1006/geno.2000.6462. PMID 11247663
- [Background] Pennarun G, Bridoux AM, Escudier E, Dastot-Le Moal F, Cacheux V, Amselem S, Duriez B. Isolation and expression of the human hPF20 gene orthologous to Chlamydomonas PF20: evaluation as a candidate for axonemal defects of respiratory cilia and sperm flagella. Am J Respir Cell Mol Biol. 2002 Mar;26(3):362-70. doi: 10.1165/ajrcmb.26.3.4738. PMID 11867345
- [Background] Omran H, Haffner K, Volkel A, Kuehr J, Ketelsen UP, Ross UH, Konietzko N, Wienker T, Brandis M, Hildebrandt F. Homozygosity mapping of a gene locus for primary ciliary dyskinesia on chromosome 5p and identification of the heavy dynein chain DNAH5 as a candidate gene. Am J Respir Cell Mol Biol. 2000 Nov;23(5):696-702. doi: 10.1165/ajrcmb.23.5.4257. PMID 11062149
- [Background] Olbrich H, Haffner K, Kispert A, Volkel A, Volz A, Sasmaz G, Reinhardt R, Hennig S, Lehrach H, Konietzko N, Zariwala M, Noone PG, Knowles M, Mitchison HM, Meeks M, Chung EM, Hildebrandt F, Sudbrak R, Omran H. Mutations in DNAH5 cause primary ciliary dyskinesia and randomization of left-right asymmetry. Nat Genet. 2002 Feb;30(2):143-4. doi: 10.1038/ng817. Epub 2002 Jan 14. PMID 11788826
- [Background] Bartoloni L, Blouin JL, Pan Y, Gehrig C, Maiti AK, Scamuffa N, Rossier C, Jorissen M, Armengot M, Meeks M, Mitchison HM, Chung EM, Delozier-Blanchet CD, Craigen WJ, Antonarakis SE. Mutations in the DNAH11 (axonemal heavy chain dynein type 11) gene cause one form of situs inversus totalis and most likely primary ciliary dyskinesia. Proc Natl Acad Sci U S A. 2002 Aug 6;99(16):10282-6. doi: 10.1073/pnas.152337699. Epub 2002 Jul 25. PMID 12142464
- [Background] Volz A, Boyle JM, Cann HM, Cottingham RW, Orr HT, Ziegler A. Report of the Second International Workshop on Human Chromosome 6. Genomics. 1994 May 15;21(2):464-72. doi: 10.1006/geno.1994.1302. No abstract available. PMID 8088851
- [Background] Meeks M, Walne A, Spiden S, Simpson H, Mussaffi-Georgy H, Hamam HD, Fehaid EL, Cheehab M, Al-Dabbagh M, Polak-Charcon S, Blau H, O'Rawe A, Mitchison HM, Gardiner RM, Chung E. A locus for primary ciliary dyskinesia maps to chromosome 19q. J Med Genet. 2000 Apr;37(4):241-4. doi: 10.1136/jmg.37.4.241. PMID 10745040
- [Background] Witt M, Wang Yf, Wang S, Sun Ce, Pawlik J, Rutkiewicz E, Zebrak J, Diehl SR. Exclusion of chromosome 7 for Kartagener syndrome but suggestion of linkage in families with other forms of primary ciliary dyskinesia. Am J Hum Genet. 1999 Jan;64(1):313-8. doi: 10.1086/302203. No abstract available. PMID 9915976
- [Background] Geremek M, Zietkiewicz E, Diehl SR, Alizadeh BZ, Wijmenga C, Witt M. Linkage analysis localises a Kartagener syndrome gene to a 3.5 cM region on chromosome 15q24-25. J Med Genet. 2006 Jan;43(1):e1. doi: 10.1136/jmg.2005.031526. PMID 16397065
- [Background] Jeganathan D, Chodhari R, Meeks M, Faeroe O, Smyth D, Nielsen K, Amirav I, Luder AS, Bisgaard H, Gardiner RM, Chung EM, Mitchison HM. Loci for primary ciliary dyskinesia map to chromosome 16p12.1-12.2 and 15q13.1-15.1 in Faroe Islands and Israeli Druze genetic isolates. J Med Genet. 2004 Mar;41(3):233-40. doi: 10.1136/jmg.2003.014084. No abstract available. PMID 14985390
- [Background] Blouin JL, Meeks M, Radhakrishna U, Sainsbury A, Gehring C, Sail GD, Bartoloni L, Dombi V, O'Rawe A, Walne A, Chung E, Afzelius BA, Armengot M, Jorissen M, Schidlow DV, van Maldergem L, Walt H, Gardiner RM, Probst D, Guerne PA, Delozier-Blanchet CD, Antonarakis SE. Primary ciliary dyskinesia: a genome-wide linkage analysis reveals extensive locus heterogeneity. Eur J Hum Genet. 2000 Feb;8(2):109-18. doi: 10.1038/sj.ejhg.5200429. PMID 10757642
- [Background] Chilvers MA, Rutman A, O'Callaghan C. Ciliary beat pattern is associated with specific ultrastructural defects in primary ciliary dyskinesia. J Allergy Clin Immunol. 2003 Sep;112(3):518-24. doi: 10.1016/s0091-6749(03)01799-8. PMID 13679810
- [Background] Rutland J, Cox T, Dewar A, Cole P. Screening for ciliary dyskinesia - a spectrum of defects of motility and structure. Eur J Respir Dis Suppl. 1983;127:71-7. PMID 6225661
- [Background] de Iongh RU, Rutland J. Ciliary defects in healthy subjects, bronchiectasis, and primary ciliary dyskinesia. Am J Respir Crit Care Med. 1995 May;151(5):1559-67. doi: 10.1164/ajrccm.151.5.7735615.
- [Background] Cazeneuve C, Ajrapetyan H, Papin S, Roudot-Thoraval F, Genevieve D, Mndjoyan E, Papazian M, Sarkisian A, Babloyan A, Boissier B, Duquesnoy P, Kouyoumdjian JC, Girodon-Boulandet E, Grateau G, Sarkisian T, Amselem S. Identification of MEFV-independent modifying genetic factors for familial Mediterranean fever. Am J Hum Genet. 2000 Nov;67(5):1136-43. doi: 10.1016/S0002-9297(07)62944-9. Epub 2000 Oct 3. PMID 11017802